CLINICAL TRIAL: NCT00696683
Title: Establishment of Natural History of Scorpion Envenomation in the Absence of Antivenom Treatment in Pediatric Patients
Brief Title: Establishment of Natural History of Scorpion Envenomation
Status: Completed | Type: Observational
Sponsor: Instituto Bioclon S.A. de C.V. (Industry)
Collaborators: University of Arizona (Other)
Responsible Party: Walter Garcia Ubbelohde MD/ Clinical Research Manager, Instituto Bioclon S.A de C.V.
Other Study IDs: AL-03/06
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Scorpion Sting Envenomation
Keywords: scorpion; sting; envenomation; antivenom
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients from the identified scorpion envenomation cases, who met inclusion/exclusion criteria.
  Interventions: Other: None, this is an observational study

INTERVENTIONS:
Other: None, this is an observational study

SUMMARY:
This retrospective study was conducted to collect data from approximately 100 patients from 6 months to 18 years of age who were stung by a scorpion but were not treated with antivenom. The study consisted of a review of hospital records of patients who were admitted for intensive care management of scorpion envenomation, at the only two hospitals in North America known to admit children routinely for scorpion sting management without antivenom. The standard of care consisted of symptomatic and supportive care, including airway maintenance, fluid and electrolyte support and, if necessary, sedation.

DETAILED DESCRIPTION:
The study objective was to document the clinical syndrome of scorpion envenomation in the absence of antivenom treatment in pediatric patients. This was done to establish historical control data on the time from sting to the time of resolution of signs of envenomation. These historical control data are intended to be used for comparison with Alacramyn treated patients in two prospective studies being conducted in Mexico and the U.S.for which a control population could not otherwise be established.

The total duration of clinically important systemic signs of envenomation was determined based upon overall investigator assessment of the last signs of any respiratory compromise, any pathological agitation or other indicator of continuing illness (e.g., continuing need for sedative administration).

To facilitate comparison of these historical data with prospective open label trials, periodic assessments of the overall presence or absence of clinically important signs was performed. Periodic assessments were also performed for each individual component indicator of respiratory compromise and of pathological agitation, when available.

A research nurse reviewed hospital discharge diagnoses for all pediatric charts coded for "scorpion sting". For these cases demographic, diagnostic, and therapeutic data were entered on the case report form (CRF) as well as data necessary to assess compliance with study inclusion and exclusion criteria.

A physician subinvestigator reviewed the research nurse's findings for the key outcome indicators, which consisted of clinically important systemic signs of scorpion envenomation and adjunctive sedation treatment (dose and timing of dose) when medical judgment was required.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 6 months to 18 years of age
* Presenting for emergency treatment with clinically important systemic signs of scorpion sting envenomation

Exclusion Criteria:

* Use of any antivenom within the last month or concomitantly
* Signs and symptoms confined to local sting site
* Concurrent medical condition involving a baseline neurologic status mimicking envenomation (chorea, tardive dyskinesia, uncontrolled epilepsy)
* Incomplete or unavailable medical record

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female patients 6 months to 18 years of age who presented for emergency treatment of scorpion sting and who had clinically important systemic signs of envenomation were included.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2004-08; Primary Completion 2004-08 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Assessment of overall duration of clinically important signs of scorpion envenomation (Clinically important signs of envenomation were divided into those indicative of respiratory distress and those comprising pathological agitation) | 4 hours or discharge

SECONDARY OUTCOMES:
To characterize treatment in the absence of antivenom (total dose, maximum rate per hour and duration of use of midazolam) | 4 hours or discharge

CONTACTS AND LOCATIONS:
Overall Officials: Walter García, MD, Study Chair — Instituto Bioclon
Locations (1):
- The University of Arizona Health Science Center & Tucson Medical Center, Tucson, Arizona, United States